CLINICAL TRIAL: NCT03569865
Title: Audio-visual Stimulation: Sleep Dose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jean Tang, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005084; 1R21NR017446-01A1 (NIH)
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Insomnia Chronic; Osteoarthritis; Pain, Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Osteoarthritis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active AVS-1 (Experimental): Active AVS-1 consists of a 30-minute pulsing lights (red, green, blue) and sounds that gradually descend from alpha (10 Hz) to delta (2 Hz).
  Interventions: Device: Audiovisual Stimulation
- Active AVS-2 (Experimental): Active AVS-2 consists of a 30-minute pulsing lights (red, green) and sounds that gradually descend from alpha (10 Hz) to delta (2 Hz).
  Interventions: Device: Audiovisual Stimulation
- Placebo AVS (Placebo Comparator): The placebo control AVS program consists of 30 minutes of constant dim light that slowly changes in color, and a steady monotone at ultra-low (<1 Hz) frequency (outside of the entrainment range).
  Interventions: Device: Audiovisual Stimulation

INTERVENTIONS:
Device: Audiovisual Stimulation — A commercially available AVS device (MindPlace Procyon) modified for use in the current study will be used to deliver the AVS programs in this study.

SUMMARY:
Osteoarthritis (OA) pain affects 50 percent of older adults, more than half of whom also experience significant sleep disturbance. This study examines the impact of an innovative audiovisual stimulation (AVS) program on human brainwaves, and its usefulness to improve sleep. The AVS intervention, if demonstrated to be efficacious for sleep promotion, could benefit millions of people worldwide.

DETAILED DESCRIPTION:
Osteoarthritis (OA) affects 50% of older adults. Common comorbidities associated with OA include poor sleep, pain, depression, and fatigue. OA patients with insomnia tend to report greater pain than those without insomnia. A recent systematic review concluded that sleep disturbance is a stronger predictor of chronic pain than vice versa. Standard treatment options for insomnia are medication and Cognitive Behavioral Therapy for Insomnia (CBT-I). Prescription medication has good short term efficacy but benefits do not persist after treatment discontinuation and there are notable side effects. Treatment effects for CBT-I are comparable to or exceed those for medications, and have been shown efficacious for persons with OA pain. However, CBT-I practitioners are not yet available in many healthcare systems. New, effective, and easy-to-use self-management alternatives could greatly help reduce the burden of insomnia and potentially decrease pain, depression, and fatigue in individuals with OA. We propose to test a novel, easily-used, self-management intervention to improve OA-related insomnia, pain, depression and fatigue: open-loop neurofeedback Audio Visual Stimulation (AVS). AVS uses preprogrammed light and sound patterns to evoke brainwave potentials at pre-set designated frequencies. The AVS intervention consists of 30 minutes of light and sound pulsing stimuli that gradually descend from alpha (10 Hz) to delta (2 Hz) frequencies. AVS placebo consists of 30 minutes of constant dim light slowly changing in color, and a steady monotone at ultra-low frequency (below 1 Hz). This proposed study builds upon our successful completion of three pilot studies using AVS. Based on the pilot findings, we hypothesize that the use of active AVS at bedtime induces delta brainwaves, but additional testing is needed to determine how long AVS should be used to produce significant improvements in subjective sleep quality relative to placebo control. In addition, we propose to experimentally test the effect of blue light, which is known to suppress melatonin production, as a potential confounding variable in the AVS intervention. We propose a trial of AVS in 75 community dwelling older adults with chronic comorbid insomnia and OA pain. After baseline assessment, participants will be randomized to 3 groups: AVS-1 (red, green & blue light) vs. AVS-2 (red & green light only) vs. placebo AVS. Participants will self-administer AVS at bedtime nightly for one month. QEEG will be measured at baseline, and then at 2, 3 and 4 weeks to evaluate neurological responses to AVS over time. Insomnia severity will be similarly assessed to determine the most efficacious AVS treatment duration and color array for improving insomnia symptoms. OA-related symptoms (pain, depression, and fatigue) and objective sleep outcomes will also be assessed. Data will inform a definitive RCT of AVS for insomnia and relative OA symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 60+ with insomnia and nonmalignant OA pain most days
* Insomnia Severity Index (ISI): >= 12
* Sleep problems >=3 times per week for >=6 months
* Brief Pain Inventory (BPI): average pain >=4 and < 10
* Osteoarthritis pain for >=6 months;
* Blessed Telephone Information-Memory-Concentration Test (TIMC) < 7
* Presence of sleep onset complaint (latency >30 minutes on PSQI OR ISI sub-scales); may also have sleep maintenance or early morning awakening complaints

Exclusion Criteria:

* Seizure disorder
* Migraine
* Photosensitivity
* Prior diagnosis of a primary sleep disorder
* Sleep apnea with an AHI/RDI score >=5 or current use of a CPAP machine
* Periodic leg movement disorder
* Restless leg syndrome
* Rapid eye movement behavior disorder
* Sleep-wake cycle disturbance
* Unusual sleep schedule (i.e. shift worker)
* 400 mg daily caffeine intake (4 cups of 8 oz brewed coffee/tea)
* 3 or more alcoholic drinks/day
* Diagnosis of: rheumatoid arthritis
* Terminal disease, pending major surgery
* Active chemotherapy or radiation for cancer
* Inpatient treatment for congestive heart failure within the previous 6 months
* Dementia diagnosis
* Use of acetylcholinesterase inhibitor and/or memantine for cognitive impairmen
* Use of psychoactive medications (stimulants, sedative hypnotics, anxiolytics, antipsychotics) or recreational drugs including marijuana.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Insomnia of Severity Index | Baseline through 4 weeks post baseline
  A 7-item questionnaire that is a global measure of perceived insomnia severity. Items use a 5-point scale for total scores of 0-28, with >15 considered moderate severity. The ISI has good internal consistency and is sensitive to changes in sleep of older adults in clinical and research.
Quantitative Electroencephalogram (QEEG) | Baseline through 4 weeks post baseline
  Cortical activity will be evaluated using a 19-channel quantitative electroencephalographic system (Discovery 24E, BrainMaster) with a standard electrode cap that has 22 sensors attaching to the scalp.

SECONDARY OUTCOMES:
Actigraphy | Baseline through 4 weeks post baseline
  Sleep and wake pattern (actigraph) will be measured by Philips Respironics Actiwatch-2. Actigraphy is a reliable and objective tool to monitor sleep-wake cycles in ambulatory individuals (including older adults) based on frequency and magnitude of movements.
Pittsburgh Sleep Quality Index (PSQI) | Baseline through 4 weeks post baseline
  Self-rating of overall sleep quality and disturbances using 7 sleep components. A PSQI global score >5 is highly sensitive and specific for distinguishing good and poor sleepers.
Brief Pain Inventory (BPI) short form | Baseline through 4 weeks post baseline
  The BPI is a 9-item questionnaire that assesses severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week.
Patient Health Questionnaire | Baseline through 4 weeks post baseline
  The PHQ-9 is a 9-item reliable, valid, measure that rates depression symptom severity on a 4-point scale.
Sleep Diary | Baseline through 4 weeks post baseline
  A 7-day diary including: bed and rise times, number of nighttime awakenings, total wake time, and morning refreshment. Participants will also report sleep and pain medication, subjective sleep quality, and pain.
Flinders Fatigue Scale | A 7-item self-report questionnaire to measure fatigue level in a variety of situations. It has strong internal reliability and validity, and been used to measure fatigue with older adults
  A 7-item self-report questionnaire to measure fatigue level in a variety of situations. It has strong internal reliability and validity, and been used to measure fatigue with older adults.
General Anxiety Disorder-7 | Baseline through 4 weeks post baseline
  A 7-item self-report questionnaire to measure anxiety level in a variety of situations.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Tang HY, Vitiello MV, Perlis M, Riegel B. Open-Loop Neurofeedback Audiovisual Stimulation: A Pilot Study of Its Potential for Sleep Induction in Older Adults. Appl Psychophysiol Biofeedback. 2015 Sep;40(3):183-8. doi: 10.1007/s10484-015-9285-x. PMID 25931250
- [Result] Tang HY, Vitiello MV, Perlis M, Mao JJ, Riegel B. A pilot study of audio-visual stimulation as a self-care treatment for insomnia in adults with insomnia and chronic pain. Appl Psychophysiol Biofeedback. 2014 Dec;39(3-4):219-25. doi: 10.1007/s10484-014-9263-8. PMID 25257144
- [Result] Tang HY, Riegel B, McCurry SM, Vitiello MV. Open-Loop Audio-Visual Stimulation (AVS): A Useful Tool for Management of Insomnia? Appl Psychophysiol Biofeedback. 2016 Mar;41(1):39-46. doi: 10.1007/s10484-015-9308-7. PMID 26294268